CLINICAL TRIAL: NCT04608461
Title: Effect of Pumpkin Seeds in the Treatment of Moderate to Severe Palmar Arsenical Keratosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Rokshana Khatun, MBBS, MD ( Phase- B ), Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2019/9986
Record Dates: First submitted 2020-10-03; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Keratotic Nodular Size

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pumpkin seeds extract containing cream (Experimental): Intervention-pumpkin seeds extract containing cream, dose-twice daily for 12 weeks
  Interventions: Drug: Pumpkin seed extract containing cream

INTERVENTIONS:
Drug: Pumpkin seed extract containing cream — Pumpkin seeds extract, white wax, white petrolium, stearyl alcohol

SUMMARY:
Arsenicosis is a major health problem in Bangladesh. Long term exposure of arsenic causes keratosis of palm which reduce working capacity of patient. It also causes massive skin lesions like Bowen's disease which has a risk to develop squamous cell carcinoma. Pumpkin seed is well known for its antioxidant and anticancer properties. So this study will be conducted to identify the compound from pumpkin seeds and to see its outcome on keratosis.

DETAILED DESCRIPTION:
Contamination of groundwater by arsenic is a global problem affecting thousands of people worldwide, especially in Bangladesh, India and West Bengal. In Bangladesh, an estimated 59 administrative districts out of 64 have been affected with significantly high concentrations of arsenic. Due to arsenicosis, keratosis of palm and sole reduce the patient's working capacity and affect the socioeconomic condition. Bowen's disease, squamous cell carcinoma and basal cell carcinoma which are invasive skin lesions also caused by arsenicosis. Keratosis can be treated by various topical preparations like salicylic acid, alpha-lipoic acid, zinc, propylene glycol, garlic oil, neem leaf extract, an extract of Azadirachta indica and Solanum melongena. But these treatments require a longer time to relieve symptoms and thus reduce patient's compliance. Pumpkin seeds are rich not only in antioxidant vitamins (carotenoids and tocopherols), minerals and proteins, but also low in fat and calories. β-carotene reduces the damage of skin from the sun and it also acts as an anti-inflammatory agent. α-carotene slows the aging process, prevents tumor growth and reduces the risk of developing cataracts. Vitamin E also called tocopherols protects the cell from oxidative damage by preventing oxidation of cell membranous unsaturated fatty acid. β-sitosterol also useful to reduce blood cholesterol and to decrease the risks of some types of cancers. So this study will be conducted to see the outcome of pumpkin seed extract in moderate to severe palmar arsenical keratosis. The study will be an open phase-II clinical trial and will be conducted in Bangabandhu Sheikh Mujib Medical University and Sirajdikhan Upazila of Munshiganj District. Extract from pumpkin seeds will be collected by using 70% ethanol as a solvent and rotary evaporator. Thin Layer Chromatography (TLC) of extract will be done to identify the compound. By using brine shrimp bioassay cytotoxicity assay will be done. The ointment will be prepared from pumpkin seeds extract and supplied to each patient at an interval of 2 weeks. Each patient will be advised about applying the cream. Improvement and adverse effects will be monitored through phone calls and during the visit regularly. Clinical improvement will be assessed by measuring the palmar arsenical nodule size before and after completion of treatment and perception of patients about their improvement. Statistical analysis and results will be documented in different diagrams and in tabulated forms.

ELIGIBILITY:
Inclusion Criteria:

* Presence of moderate to severe palmar arsenical keratosis
* Drinking arsenic contaminated water for at least six months
* Patient voluntarily agreed to participate

Exclusion Criteria:

* Age less than 19 years or more than 65 years
* Pregnant and nursing mother
* Skin diseases like atopic dermatitis eczema and psoriasis

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
Keratotic nodular size | 12 weeks
  Nodular size and lesion size will be measured by slide calipers

CONTACTS AND LOCATIONS:
Locations (1):
- Sirajdikhan, Munshiganj, Bangladesh

IPD SHARING:
Plan to Share IPD: No